CLINICAL TRIAL: NCT06229756
Title: Clinical Results of Asqelio™ EDOF Toric Soft Hydrophobic Intraocular Lens After Cataract Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: AST Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ASQE012022
Record Dates: First submitted 2024-01-18; First posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EDOF Toric: Patient submitted to bilateral implantation of Asqelio EDOF Toric IOL

SUMMARY:
The goal of this observational study is to assess the clinical outcomes of binocular implantation of Asqelio EDOF Toric IOLs in healthy cataract patients. The main questions it aims to answer are:

* What is the visual performance at different distances 3 months after implantation of Asqelio EDOF Toric in both eyes?
* What is the amount of residual refractive error following the implantation?
* What is the contrast sensitivity of patients 3 months after implantation of Asqelio EDOF Toric in both eyes?
* What is the optical quality of the eye implanted with Asqelio EDOF Toric IOL?
* What is the incidence and severity of visual symptoms after implantation of Asqelio EDOF Toric?
* What is the level of patient satisfaction after implantation of Asqelio EDOF Toric?

For this purpose, participants will be submitted to a comprehensive visual and refractive assessment, following common clinical practice, 3 months after binocular implantation of Asqelio EDOF Toric IOLs, and asked to complete visual symptoms and patient satisfaction questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Patients 50 years old or more submitted to bilateral cataract surgery and implanted with Asqelio EDOF toric IOL, with cylinder value of 0.0 D.
* Patients signing informed consent
* Transparent media except for the cataracts
* Potential postoperatoria visual acuity of 20/25 or better

Exclusion Criteria:

* Preoperative corneal astigmatism greater than 1.00D
* Patients who do not provide informed consent
* Patients who do not understand the study procedure
* Previous corneal surgery or trauma
* Irregular cornea (e.g. keratoconus)
* Choroidal hemorrhage
* Microphtalmos
* Severe corneal dystrophy
* Uncontrolled or medically controlled glaucoma
* Clinically significant macular changes
* Concomitant severe eye disease
* Non-age-related cataract
* Severe optic nerve atrophy
* Diabetic retinopathy
* Proliferative diabetic retinopathy
* Amblyopia
* Extremely shallow anterior camera
* Severe chronic uveítis
* Pregnant or nursing
* Rubella
* Mature/dense cataract that makes it difficult to examine the fundus preoperatively.
* Previous retinal detachment
* Concurrent participation in other research with drugs or clinical devices
* Expect to require another eye surgery during the study period

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects submitted to bilateral cataract surgery with implantation of extended depth of focus IOLs according to common clinical practice
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-10-26 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Uncorrected Monocular Visual acuity for distance | 3 months after implantation
  Visual acuity without additional correction determined at a distance of 4 m in LogMAR units
Uncorrected Monocular Visual acuity for intermediate distance | 3 months after implantation
  Visual acuity without additional correction determined at a distance of 67 cm in LogMAR units
Uncorrected Monocular Visual acuity for near distance | 3 months after implantation
  Visual acuity without additional correction determined at a distance of 40 cm in LogMAR units
Corrected Monocular Visual acuity for distance | 3 months after implantation
  Visual acuity with best correction determined at a distance of 4 m in LogMAR units
Corrected Monocular Visual acuity for intermediate distance | 3 months after implantation
  Visual acuity with best correction determined at a distance of 67 cm in LogMAR units
Corrected Monocular Visual acuity for near distance | 3 months after implantation
  Visual acuity with best correction determined at a distance of 40 cm in LogMAR units
Refractive error | 3 months after implantation
  Residual refractive error after implantation obtained by subjective refraction methods

SECONDARY OUTCOMES:
Contrast sensitivity function under photopic conditions | 3 months after implantation
  Contrast sensitivity measured under photopic conditions for spatial frequencies of 3, 6, 12 and 18 cycles per degree using the Clinical Trial Suite in logCS units
Contrast sensitivity function under mesopic conditions | 3 months after implantation
  Contrast sensitivity measured under mesopic conditions for spatial frequencies of 1.5, 3, 6 and 12 cycles per degree using the Clinical Trial Suite in logCS units
Contrast sensitivity function under photopic conditions with glare | 3 months after implantation
  Contrast sensitivity measured under photopic conditions inducing glare, for spatial frequencies of 3, 6, 12 and 18 cycles per degree using the Clinical Trial Suite in logCS units
Contrast sensitivity function under mesopic conditions with glare | 3 months after implantation
  Contrast sensitivity measured under mesopic conditions inducing glare, for spatial frequencies of 1.5, 3, 6 and 12 cycles per degree using the Clinical Trial Suite in logCS units
Binocular defocus curve | 3 months after implantation
  Visual acuity in logMAR units under binocular conditions, determined varying the stimulus mergence using lenses from -4.00D to +2.00D in 0.50D steps and best refractive correction for distance
Aberrometry | 3 months after implantation
  Optical quality measured as Zernike coefficients for total Root Mean Square of Higher order aberrations, and Spherical aberrations, expressed in microns
Light distortion | 3 months after implantation
  Distortion of light as light distortion index, determined by means of the light distortion analyzer
Patient-reported visual symptoms | 3 months after implantation
  Incidence and severity of visual symptoms, determined by means of a visual symptoms questionnaire. Incidence will be scored in a scale from 1 (never) to 4 (always), severity from 1 (none) to 4 (severe), and bothersome rom 1(none) to 4 (a lot)
Patient-reported satisfaction | 3 months after surgery
  Level of satisfaction with vision and difficulty performing daily activities, determined by means of the CATQuest 9SF questionnaire, where items are scored in a scale from 1 (yes, a lot of difficulties) to 4 (no, no difficulties) and a "cannot decide" option. Satisfaction is scored from 1 (very unsatisfied) 4 (very satisfied) and a "cannot decide" option
Incidence of Adverse events | 3 months after surgery
  Percentage of patients presenting adverse events (ocular and non ocular, severe and not severe), including secondary surgical procedures

CONTACTS AND LOCATIONS:
Locations (1):
- OftalVist Alicante, Alicante, Spain